CLINICAL TRIAL: NCT04362150
Title: Long-term Impact of Infection With Novel Coronavirus (LIINC): An Observational Study
Brief Title: Long-term Impact of Infection With Novel Coronavirus (COVID-19)
Acronym: LIINC
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 20-30479
Record Dates: First submitted 2020-04-23; First posted 2020-04-24 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: COVID
Keywords: COVID-19; coronavirus; SARS-CoV-2; Long COVID; post-acute sequelae of SARS-CoV-2
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, peripheral blood mononuclear cells, plasma, serum, and saliva.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 positive, recovered: Individuals with positive test for COVID-19 who have recovered from acute infection (21 days after symptom onset + improvement in symptoms + resolution of fever for 72 hours without fever reducing medicines).

SUMMARY:
LIINC is a study of volunteers who were previously infected with SARS-CoV-2 (also known as novel coronavirus or COVID-19) who have recovered from acute infection. The study is designed to provide a specimen bank of samples with carefully characterized clinical data. LIINC specimens will be used to examine multiple questions involving the virologic, immunologic, and host factors involved in COVID-19, with a focus on understanding variability in the long-term immune response between individuals.

DETAILED DESCRIPTION:
LIINC is an observational, prospective study of individuals previously infected with SARS-CoV-2 who have recovered from acute illness. The overall objective of the study is to investigate the clinical consequences of SARS-CoV-2 infection. These include the pre-existence and development of medical conditions, measures of immune activation and inflammation, changes in immunologic function, and variability in host responses. There will be a specific focus on demographic differences including age, gender, and race.

Enrolled volunteers are seen at San Francisco General Hospital at baseline, monthly for 3 months and then every 3 months for up to 2 years. Visits include a detailed interview, saliva collection, and a blood draw. Baseline visits take approximately 90 minutes, and follow up visits take approximately 20-40 minutes. No personal identifiers are used for specimen bank samples.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent, and
2. Age >/= 18 years, and
3. A history of SARS-CoV-2 infection, as evidenced by:

   1. Available laboratory documentation of SARS-CoV-2 RNA positivity on a nucleic acid amplification test or by serologic testing when this becomes available, or
   2. Reference by the participant to a laboratory test performed on respiratory tract secretions or blood, fingerstick, or saliva test that was reported to the participant to be positive for SARS-CoV-2 or COVID-19 infection,
4. And a period of 21 days or more has elapsed since the first positive test or symptoms preceding the first positive test, whichever is earlier.

Exclusion Criteria:

1. Self-reported or documented chronic anemia with hemoglobin < 9 g/dL. Anemia during a preceding acute illness will not be exclusionary.
2. Serious medical or psychiatric illness that, in the opinion of the site investigator, would interfere with the ability to adhere to study requirements or to give informed consent.
3. Active drug or alcohol use or dependence that, in the opinion of the Principal Investigator, would interfere with adherence to study requirements or to give informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will enroll individuals with prior SARS-CoV-2 infection across a wide spectrum of age, race, gender, and disease severity.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2020-04-21 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Participant age | Baseline visit
  The median age of study participants at enrollment.
Participant sex | Baseline visit
  The proportion of men and women participating in the baseline visit.
Participant race/ethnicity | Baseline visit
  The proportion of participants from each demographic group.
Proportion of participants previously hospitalized. | Baseline visit
  The proportion of participants who were previously hospitalized.

SECONDARY OUTCOMES:
Long COVID Outcomes | 4, 8, 12, 16, 20, and 24 months post-COVID.
  The proportion of participants meeting various case definitions of Long COVID.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Deeks, MD, Principal Investigator — University of California, San Francisco; Michael J Peluso, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital (ZSFG), San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peluso MJ, Deveau TM, Munter SE, Ryder D, Buck A, Beck-Engeser G, Chan F, Lu S, Goldberg SA, Hoh R, Tai V, Torres L, Iyer NS, Deswal M, Ngo LH, Buitrago M, Rodriguez A, Chen JY, Yee BC, Chenna A, Winslow JW, Petropoulos CJ, Deitchman AN, Hellmuth J, Spinelli MA, Durstenfeld MS, Hsue PY, Kelly JD, Martin JN, Deeks SG, Hunt PW, Henrich TJ. Chronic viral coinfections differentially affect the likelihood of developing long COVID. J Clin Invest. 2023 Feb 1;133(3):e163669. doi: 10.1172/JCI163669. PMID 36454631
- See also: Long-term Impact of Infection with Novel Coronavirus study website — https://www.liincstudy.org/en/home